CLINICAL TRIAL: NCT07367802
Title: Exploring the Benefits of a 3D Patient-specific Alignment in Total Knee Arthroplasty
Acronym: iKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, zhijun li, KUleuven Brugge, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S67874; B3222022001251 (Other: Ethics Committee Research UZ/KU Leuven)
Record Dates: First submitted 2025-12-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: TKA Outcomes
Keywords: TKA; iKA; aMA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To examine the lower limb kinematic differences during the challenging daily functional movements, s (Experimental): To examine the lower limb kinematic differences during the challenging daily functional movements, such as the lunge, in individuals who have undergone iKA TKA, compared to those with aMA TKA and healthy controls.
  Interventions: Procedure: iKA

INTERVENTIONS:
Procedure: iKA — This study compared inverse kinematic alignment (iKA) TKA, which preserves native JLO, with adjusted mechanical alignment (aMA) TKA, which standardizes JLO to 90°, and a healthy control group across eight functional activities.

SUMMARY:
General Aim: to explore the iKA in TKA related to clinical, biomechanical, and functional outcomes.

DETAILED DESCRIPTION:
First specific aim: to investigate the kinematics during daily functional movements in individuals with the iKA TKA to those with aMA TKA, as well as the healthy control group.

Second specific aim: to investigate kinetics and muscle activation patterns during functional movements in individuals with the iKA aligned TKA to those with aMA TKA, as well as a healthy control group.

Third specific aim: to investigate the impact of the whole body on functional outcomes following iKA and aMA TKA, in comparison to the healthy control group, and to explore the underlying factors contributing to suboptimal outcomes.

ELIGIBILITY:
Inclusion Criteria:

were age under 85 years. primary robot-assisted TKA using either iKA or aMA. surgery performed two years before enrollment. independent ambulation without assistive devices; and informed consent.

Exclusion Criteria:

history of lower limb trauma or fracture. neurological disorders (e.g., stroke, Parkinson's disease, multiple sclerosis). systemic musculoskeletal diseases (e.g., rheumatoid arthritis, diabetic neuropathy).

revision arthroplasty. and cognitive impairment affecting study participation.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Height | 2 years after TKA
  Stadiometer; height in millimeters
Joint angles | 2 years after surgery
  Vicon Nexus 2.12 software (©Vicon Motion Systems Ltd., Oxford, UK); Unit: Degrees
Age | 2 years after TKA
  year
Leg Length | 2 years after TKA
  Direct Tape Measure; Leg Length in millimeters
Inter-ASIS Dist | 2 years after TKA
  Vernier caliper， Inter-ASIS Dist in millimeters
Knee Width | 2 years after TKA
  Vernier caliper, Knee Width in millimeters
Ankle Width | 2 years after TKA
  Vernier caliper, Ankle Width in millimeters
Elbow Width | 2 years after TKA
  Vernier caliper, Elbow Width in millimeters
Wrist Width | 2 years after TKA
  Vernier caliper, Wrist Width in millimeters
Hand Thickness | 2 years after TKA
  Vernier caliper, Hand Thickness in millimeters
Total Gait Cycle Duration | 2 years after TKA
  Vicon Nexus 2.12 software (©Vicon Motion Systems Ltd., Oxford, UK); Unit in second
Visual Analog Scale | Pre-TKA, 6 weeks after TKA, 2 years after TKA
  Pain Scores
Oxford Knee Score (OKS) | Pre-TKA; 2 years after TKA
  total score ranging from 0 to 48
maximum voluntary isometric strength tests of the lower limb | 2 years after TKA
  Peak force measured with a hand-held dynamometer (Micro FET 2 Handheld Dynamometer, Hoggan, USA); Unit: Newtons
Muscle activity patterns for eight muscles (gluteus medius, rectus femoris, vastus medialis, vastus lateralis, biceps femoris, semitendinosus, tibialis anterior and gastrocnemius medialis) | 2 years after TKA
  A 16-channel telemetric wireless surface electromyography (EMG) system (Waveplus®, Cometa, Rome, Italy) operating at 1000 Hz was utilized. Unit: Volt

SECONDARY OUTCOMES:
BMI | 2 years after TKA
  weight and height will be combined to report BMI in kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Bruges, West, Belgium

IPD SHARING:
Plan to Share IPD: No
it is a 15 year study

REFERENCES:
- [Result] Winnock de Grave P, Kellens J, Luyckx T, Tampere T, Lacaze F, Claeys K. Inverse Kinematic Alignment for Total Knee Arthroplasty. Orthop Traumatol Surg Res. 2022 Sep;108(5):103305. doi: 10.1016/j.otsr.2022.103305. Epub 2022 May 2. PMID 35513224

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT07367802/Prot_SAP_000.pdf